CLINICAL TRIAL: NCT06428552
Title: To Evaluate the Efficacy of Mobile Applications in Tailoring and Enhancing Rehabilitation Interventions for Pediatric Patients With Cerebral Palsy
Brief Title: To Evaluate the Efficacy of Mobile Applications in Tailoring and Enhancing Rehabilitation Interventions for Pediatric CP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSRSW/Batch-Fall22/712
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual care at home for 12 weeks (Experimental): Daily rehabilitation program of 40 minutes duration using a mobile application to be completed 6 days per week for 12 weeks
  Interventions: Device: Mobile Application

INTERVENTIONS:
Device: Mobile Application — Daily rehabilitation program of 40 minutes duration using a mobile application to be completed 6 days per week for 12 weeks

SUMMARY:
The world of technology is changing and becoming more advanced. Children with cerebral palsy can benefit from the technology to enhance their mobility, balance, and coordination through mobile applications. A lot of applications are made to offer games and interactive therapy activities that focus on balance, coordination, and motor skills.

DETAILED DESCRIPTION:
They may find these activities entertaining as well as helpful, which makes their rehabilitation more pleasurable. This work builds on previous studies by making a mobile application that may be accessed from any location, giving therapeutic treatments more distribution flexibility. This is especially helpful for those with cerebral palsy who might have mobility issues that make it challenging to consistently attend in-person therapy sessions. Cerebral palsy children can perform organized exercises at home with the help of mobile application made for therapeutic activities and rehabilitation. Therapeutic activities may be customized to meet the unique demands of each patient, guaranteeing that the treatment plan is in line with their capabilities and objectives. Caregiver's involvement in the treatment process is a common element of app created specifically for people with cerebral palsy. This might involve providing tools to enhance home-based care, educating caregivers through resources, and monitoring progress in order to promote a team-based approach to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy
* Children aged between 5 to 16 years

Exclusion Criteria:

* Children with unstable epilepsy, chronic heart abnormalities , asthma , anemia and other medical conditions
* undergone botulinum neurotoxin A (BoNT-A)injections or surgery in the previous 2 months or 6 months respectively. "

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
questionnaire(QUIS)the application software | 12 Months
  questionnaire(QUIS)the application software has been given to the intervention group and after using the software for one week, all participants answered the user satisfaction interaction questionnaire(QUIS).This step has taken to assess the software's usability based on feedback taken from parents or caregivers of patient with cerebral palsy and to assess the impact of utilizing this mobile application.
Pedi Cat Questionnaire | 12 months
  Pedi Cat Questionnaire To assess amount of recovery in patients with cerebral palsy, the intervention group answered valid and reliable Pedi Cat questionnaire at the first day of the study. The intervention group used the content and rehabilitation protocol of the app under the supervision of therapist for 12 weeks at home. After 12 weeks, the Pedi Cat questionnaire was answered by intervention group to assess recovery increasing or any change in the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Hope Rehabilitaion Centre, Mansoor Hospital Lahore , ChildRehab Sangla Hill, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No